CLINICAL TRIAL: NCT01345266
Title: Characterisation of Healthy Volunteers, Asthma and Chronic Obstructive Pulmonary Disease Patients for Inhalation Profile, Pharyngometry, Spirometric Indices and Lung Morphometry
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 113817
Record Dates: First submitted 2010-10-07; First posted 2011-05-02 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pharyngometry; Novel Dry Powder Inhaler; HRCT; Inhalation Profiles
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inhalation Profiling (Other): All subjects have Inhaltion profiling, there are no other arms.
  Interventions: Procedure: Inhalation Profiling

INTERVENTIONS:
Procedure: Inhalation Profiling — All subects recieve Inhaltion Profiling there are no interventions.

SUMMARY:
This is a clinical study, with no investigational product, to characterise the inhalation profiles of healthy volunteers, volunteers with mild, moderate and severe Asthma and volunteers with mild, moderate and severe Chronic Obstructive Pulmonary Disease (COPD), through the novel dry powder inhaler.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply.

* All volunteers must be aged between 21 to 70 years inclusive and be competent to understand and give informed consent.
* All female volunteers of child bearing potential must have provided a negative pregnancy test before inclusion and prior to any HRCT scan.
* Body weight < 120 kg and BMI within the range 18 - 35 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete the study
* Subject will then be included only if they fulfil all criteria for the following relevant cohort Healthy: Cohort
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history and physical. A subject with a clinical abnormality or parameters outside the reference range for the population being studied may be included if the Investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Non-smokers (never smoked or not smoking for >12 months with <1 pack year history) (Pack years = (cigarettes per day smoked/20) x number of years smoked))
* No history of a chronic respiratory disorder.
* No history of acute respiratory disease within four weeks prior to inclusion.
* No history of breathing problems such as a history of asthma, unless the asthma was in childhood and has now completely resolved, no longer requiring maintenance or intermittent therapy.
* No other significant medical disorder that may affect the respiratory system or that causes significant disability.

Asthmatic: Cohort

* Clinically diagnosed with asthma, for at least 6 months, stratified as either: mild, moderate or severe, based on current treatment, using the British Thoracic Society - - Guidelines on Asthma [BTS, 2009]. For inhaled steroid equivalence to budesonide please refer to the GINA guidelines [GINA, 2008]
* Mild, defined Step 1 or 2 by BTS Asthma Guidelines
* Moderate, defined as step 3 by BTS Asthma Guidelines
* Severe, defined as step 4 or 5 by BTS Asthma Guidelines
* Non-smokers (never smoked or not smoking for >12 months with <1 pack year history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
* Able to withhold from short acting bronchodilators for 6 hours and long acting bronchodilators for 12 hours before study assessments
* No history of acute respiratory disease within four weeks prior to inclusion.
* No history of any other inflammatory lung condition or carcinoma of the lung.
* No exacerbation of disease requiring hospitalisation within previous four weeks.

COPD: Cohort

- Clinically diagnosed COPD, for at least 6 months prior to screening, either: mild, moderate or severe/very severe (stage I, II, III/IV) COPD as defined by GOLD guidelines [GOLD 2008]. The following lung function criteria are post bronchodilator

Stage I:

* Mild COPD. FEV1/FVC < 70%, FEV1 ≥ 80% predicted with or without chronic symptoms (cough, sputum production) Stage II
* Moderate COPD. FEV1/FVC < 70%. 50% ≤ FEV1 < 80% predicted with or without chronic symptoms (cough, sputum production) Stage III and IV
* Severe COPD. FEV1/FVC < 70%. 30% ≤ FEV1 < 50% predicted with or without chronic symptoms (cough, sputum production)
* Very Severe COPD.FEV1/FVC < 70%, FEV1 < 30% predicted or FEV1 < 50% predicted plus chronic respiratory failure
* Subject is a smoker or an ex-smoker with a smoking history of at least 10 pack years (Pack years = (cigarettes per day smoked/20) x number of years smoked)).
* No history of acute respiratory disease within four weeks prior to inclusion
* No history of any other inflammatory lung condition or carcinoma of the lung.
* No exacerbation of disease requiring hospitalisation within previous four weeks.
* Able to withhold from short acting bronchodilators for 6 hours and long acting bronchodilators for 12 hours before study assessments

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* As a result of the medical interview, physical examination or screening investigations, the physician responsible considers the volunteer unfit for the study.
* Any pregnant female
* Volunteers who have a past or present disease, which as judged by the Investigator, may affect subject safety or influence the outcome of the study.
* The subject has received an investigational drug or participated in any other research trial within 30 days or five half-lives, or twice the duration of the biological effect of any drug (whichever is longer).
* The subject that has both asthma and COPD.
* Previous inclusion in a research and/or medical protocol involving nuclear medicine,
* Any Radiological investigations with significant radiation burden (a significant radiation burden being defined as ICRP category IIb or above: No more than 10 mSv in addition to natural background radiation, in the previous 3 years including the dose from this study).
* The subject has a history of alcohol or drug abuse.
* The subject has had a respiratory tract infection within four weeks of the start of the study.
* The subject has a history of claustrophobia.
* The subject is unable to perform the Multi Channel Recorder and/or Pharyngometry assessments correctly.
* The subject has a known allergy or hypersensitivity to milk protein.
* Unwillingness or inability to follow any of the procedures outlined in the protocol.
* Subject is kept under regulatory of judicial order in an institution.
* Subject is mentally or legally incapacitated.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-06-28 (Actual); Study Completion 2010-06-28 (Actual)

PRIMARY OUTCOMES:
Inhaltion Profile Recording (IPR): Measures will be Peak Pressure Drop (kPa), Peak Inspiratory Flow Rate (L/min), Inhaled Volume (L), Inhalation time (s) Average Inhalation flow rate (L/min) | 24 hours
  To characterise the inhalation profiles of healthy volunteers, volunteers with mild, moderate and severe asthma and volunteers with mild, moderate and severe COPD, through the novel DPI, using the IPR
Pharangometry: Measures will be, Distance (cm) Volume (cm3) Average cross sectional area (cm2) | 24 hours
  To characterise the inhalation profiles of healthy volunteers, volunteers with mild, moderate and severe asthma and volunteers with mild, moderate and severe COPD, using pharangometry

SECONDARY OUTCOMES:
HRCT scans: Measures are Total Lung Capacity (TLC) and Functional Residual capacity (FRC) | 24 hours
  Exploratory: To provide data from HRCT scans, spirometry and plethysmography measures which will enable further work in the mapping of the small and large airways and deliver 3D geometries of these airways.
Lung function indices by spirometry: Measures, FEV1, Vmax25 and 50, PEFR, PIFR | 24 hours
  Exploratory: To provide data from HRCT scans, spirometry and plethysmography measures which will enable further work in the mapping of the small and large airways and deliver 3D geometries of these airways.
Whole body plethysmography: Measures include.Volume: total lung, residual volume, functional reserve volume, Impedance - generation 0 to 6, Resistance - generation 0 to 6 and Diffusion. | 24 hours
  Exploratory: To provide data from HRCT scans, spirometry and plethysmography measures which will enable further work in the mapping of the small and large airways and deliver 3D geometries of these airways.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Belgium (2):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Edegem

REFERENCES:
- [Derived] Prime D, de Backer W, Hamilton M, Cahn A, Preece A, Kelleher D, Baines A, Moore A, Brealey N, Moynihan J. Effect of Disease Severity in Asthma and Chronic Obstructive Pulmonary Disease on Inhaler-Specific Inhalation Profiles Through the ELLIPTA(R) Dry Powder Inhaler. J Aerosol Med Pulm Drug Deliv. 2015 Dec;28(6):486-97. doi: 10.1089/jamp.2015.1224. Epub 2015 Sep 15. PMID 26372467
- [Derived] Hamilton M, Leggett R, Pang C, Charles S, Gillett B, Prime D. In Vitro Dosing Performance of the ELLIPTA(R) Dry Powder Inhaler Using Asthma and COPD Patient Inhalation Profiles Replicated with the Electronic Lung (eLung). J Aerosol Med Pulm Drug Deliv. 2015 Dec;28(6):498-506. doi: 10.1089/jamp.2015.1225. Epub 2015 Sep 15. PMID 26372465
- See also: Results for study 113817 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113817?search=study&study_ids=113817#rs